CLINICAL TRIAL: NCT03286790
Title: Incidence of pNeumonia and Related ConseqUences in Nursing Home
Brief Title: Incidence of pNeumonia and Related ConseqUences in Nursing Home Residents
Acronym: INCUR
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: 11 280 03
Record Dates: First submitted 2017-09-14; First posted 2017-09-18 (Actual); Last update posted 2017-09-18 (Actual); Status verified 2017-09

CONDITIONS: Pneumonia
Keywords: elderly
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Data collection on pneumonia events

SUMMARY:
In the present proposal, we hypothesize that specifically targeting pneumonia events with preventive interventions in the French EHPAD (Etablissements d'Hébergement pour Personnes Agées Dépendantes) setting (thus, improving the health status and quality of life of patients) may simultaneously produce relevant reductions in the healthcare costs. In fact, although the number of pneumonia cases may be numerically limited, the consequences of each event are potentially catastrophic for both the patient and the healthcare system. Unfortunately, to date, information about the incidence and economical effects of pneumonia in the older population living in the French EHPAD are extremely scare. To adequately evaluate whether there is room to implement preventive interventions aimed at reducing the onset of pneumonia in a cost-effective fashion on a large scale, preliminary data from this specific population are needed. This first step is crucial towards the appropriate design and conduction of possible future large-scale intervention trials in the EHPAD setting.

ELIGIBILITY:
Inclusion Criteria:

* Groups Iso-Resources (GIR) ranging between 5 (included) and 2 (included)
* Ability and willingness to participate to the study and to provide informed consent
* Agreement with the patient's physician about the enrolment to the study

Exclusion Criteria:

* Refusal of the EHPAD to participate
* Patients with severe disability (GIR 1)
* Patients with no evidence of functional impairment (GIR 6)
* Patients living in the participating EHPAD for less than 30 days since the baseline study visit

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients living in the participating EHPAD for more than 30 days since the baseline study visit
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Incidence of pneumonia | months 12
  Estimate the incidence of pneumonia events in a sample of 800 older patients living in 30 EHPADs over a period of 12 months
healthcare costs | months 12
  To compare the healthcare costs of participants experiencing a pneumonia event versus those who will not in a random sample of 800 older patients living in 30 EHPADs over a period of 12 month

SECONDARY OUTCOMES:
Mortality risk | Months 12
  To calculate the mortality risk in a random sample of 800 EHPAD older patients according to the presence/absence of a pneumonia event occurred during a follow-up period of 12 months
Physical Function | Months 12
  To measure the physical function modifications experienced by a random sample of 800 EHPAD older patients according to the presence/absence of a pneumonia event occurred during a follow-up period of 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Mateo Cesari, MD, Study Director — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No